CLINICAL TRIAL: NCT02993913
Title: A Safety, Tolerability and Pharmacokinetic Study of Single and Repeat Oral Escalating Doses of Simmiparib in Patients With Advanced Malignant Tumors
Brief Title: Safety, Tolerability and Pharmacokinetics of Simmiparib in Patients With Malignant Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Acebright Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ACE-CT-006I
Record Dates: First submitted 2016-12-06; First posted 2016-12-15 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-12

CONDITIONS: Malignant Advanced Solid Tumor
MeSH Terms: interventions — simmiparib

ARMS (1):
- Simmiparib tablet monotherapy (Experimental): Drug: Simmiparib tablet oral Qd or Bid
  Interventions: Drug: Simmiparib

INTERVENTIONS:
Drug: Simmiparib — Simmiparib Tablets, oral administration
  Other Names: SMOCL-9112

SUMMARY:
Phase I dose escalating trial. Primary objectives of this study are to assess the safety and tolerability of Simmiparib following single and multiple oral doses in patients with advanced solid malignancies, to determine the maximum tolerance dose (MTD) and dose limiting toxicity (DLT), and pharmacokinetic profile.

The Secondary objective is to observe the preliminary antitumor effect of Simmiparib.

DETAILED DESCRIPTION:
This single-center, nonrandomized, open-label, dose-escalating study. The trial was divided into dose escalation and expansion stages.

ELIGIBILITY:
Inclusion Criteria:

1. Patients confirmed with advanced solid tumor based on pathology and/or cytology, considered unresponsive or poorly responsive to standard therapies, no curative therapies or can't tolerate standard therapies;
2. Patients must have measurable disease in accordance with RECIST criteria v. 1.1, at least one lesion that can be accurately measured in CT and MRI at least one dimension ( longest diameter≥10mm; if lymph node, short diameter≥15mm );
3. Age≥18 and ≤75 years, both men and women, no history of drug abuse and alcohol;
4. Life expectancy≥ 3 months and can be followed for safety and efficiency
5. Received no prior anti-tumor therapies at least within past 4 weeks and no other adjuvant anti-tumor regimen(including steroids mediations )
6. Have recovered to≤ common terminology criteria of adverse events (CTC-AE) 1 from toxicities of prior therapy
7. Not participated in any clinical trials within 28 days;
8. Not have received treatment of poly-ADP ribose polymerase (PARP) inhibitor;
9. No serious abnormal hematopoiesis function, has adequate cardiac, pulmonic, hepatic and renal function. Blood routine and blood biochemical examination within 2 weeks before enrollment : White blood cell (WBC) ≥4000/mm3, Absolute neutrophil count (ANC) ≥1,500/mm3, Platelets ≥100,000/mm3, Coagulation function ≤ 1.5 times upper limit of normal (ULN), serum creatinine ≤ 1.5 times ULN, Total bilirubin ≤ 1.5 times ULN, Patients without liver metastasis, Aspartate aminotransferase (AST)/alanine aminotransferase (ALT)≤ 2.5 times ULN; Patients with liver metastasis, Aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/≤ 2.5 times ULN, NYHAclass≤Ⅱand Left ventricular ejection fraction ( LVEF)>50%;
10. Virology test: negative HbsAg, HCV, HIV and syphilis
11. Eastern Cooperative Oncology Group(ECOG) performance status ≤2;
12. No history of other malignant tumors, except cervical carcinoma in situ, basal skin cancer or squamous-cell carcinoma that have been cured; No other serious illnesses that are in conflict with this study and significant heart disease and psychosis;
13. Ability to understand and a willingness to sign a written informed consent; Obtaining consent before any operation

Exclusion Criteria:

1. Patients with serious medical disease, including, severe cardiopathy, vascular disease, uncontrolled diabetes, uncontrolled hypertension, severe infection , or psychosis, etc.;
2. Patients with primary brain lesion or metastases lesion;
3. Female patient who is pregnant, breast feeding or unwilling to contraception;
4. Patient who received or is receiving any other investigational agents within 4 weeks prior to treatment;
5. Patients, with poor compliance, or based on the opinion of the investigator, should not be enrolled into this study;
6. has not recovered to grade 1 or better from any adverse events related to previous therapy.
7. Neurotoxicity observed in previous antineoplastic therapy has not recovered to grade 1 or below.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Per doselevel of 3 to 6 patients (When 3-6 patients have completed DLT periods of 4 weeks)
  The Dose level at which more than 1/6 patients develop a Dose Limiting Toxicity (DLT)
Pharmacokinetic Cmax (maximum concentration) | At day 1 single dose period, day 8 and 28 multiple dose period day
  PK blood collection Before 0:00h and after 0.25h、0.50h、1:00h、1.50h、2:00h、3:00h、4:00h、6:00h、8:00h、10:00h、24:00h、48:00h、72:00h at single dose period.
  PK blood collection before 0:00h and after 0.25h、0.50、1:00h、1.50h、2:00h、3:00h、4:00h、6:00h、8:00h、10:00h and 12:00h at multiple dose period
Pharmacokinetic Tmax (Time of maximum concentration) | At day 1 single dose period, day 8 and 28 multiple dose period day
Pharmacokinetics AUC (Area Under the Curve) | At day 1 single dose period, day 8 and 28 multiple dose period day

SECONDARY OUTCOMES:
Poly ADP-ribose polymerase (PARP) inhibition measured by PAR assay | Up to 4 months
Overall Response Rate (ORR) | Up to 4 months
  ORR according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China